CLINICAL TRIAL: NCT01752595
Title: The Music Activity INTervention for Adherence Improvement Through Neurological Entrainment Study
Brief Title: The Music Activity INTervention for Adherence Improvement Through Neurological Entrainment
Acronym: MAINTAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Ontario Centres of Excellence (Industry); University of Toronto (Other)
Responsible Party: Principal Investigator, Dr. David Alter, Dr. David Alter, MD, PhD, FRCPC, Toronto Rehabilitation Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-035
Record Dates: First submitted 2012-12-03; First posted 2012-12-19 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Myocardial Infarction; Compliance Behavior; Patient Compliance
MeSH Terms: conditions — Myocardial Infarction; Patient Compliance

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Standard (No Intervention): Subjects randomized to this group will receive standard, usual care with no intervention.
- Preference Based Music Intervention (Active Comparator): Subjects randomized to this arm will receive an iPod player and an activity monitoring device. The iPod will be loaded with patient indicated music preferences that is synched to the patients pace prescription. Subjects will be asked to use their iPod player during off-site exercise periods.
  Interventions: Other: Preference Based Music Intervention
- Preference Based Rhythmic Auditory Stimulation Music (Active Comparator): Subjects randomized to this arm will receive an iPod player and an activity monitoring device. The iPod will be loaded with patient indicated music preferences that is synched to the patients pace prescription. Subjects will be asked to use their iPod player during off-site exercise periods. Rhythmic Auditory Stimulation (accentuation of beats, frequencies) will be added to the music subliminally.
  Interventions: Behavioral: Preference Based Rhythmic Auditory Stimulation Music

INTERVENTIONS:
Behavioral: Preference Based Rhythmic Auditory Stimulation Music — Patients that have been randomized into arms 2 and 3 will be blinded to the intervention they are receiving (i.e. preference-based playlist vs. preference-based playlist that has been edited to include Rhythmic Auditory Stimulation (RAS). RAS drives synchronous neural oscillation (entrainment) and functions in two ways: (1) facilitates pace and heart-rate synchrony and (2) facilitates brain state dominance (getting into the zone). RAS will be accomplished through: (1) sequencing of subject self-selected music based on tempo, (2) accentuation of the rhythmic driving pulse with added percussive-type sounds, (3) addition of binaurally detuned pitches to follow bass lines at brain-state target frequencies (e.g., 8 Hz alpha, or 16 Hz beta), and (4) the addition of binaurally detuned "background" sounds (e.g., low frequency hum) at target Hz frequencies. RAS is implemented as inherent and natural to the music and may remain imperceptible to most.
  Arms: Preference Based Rhythmic Auditory Stimulation Music
Other: Preference Based Music Intervention
  Arms: Preference Based Music Intervention

SUMMARY:
Auditory motor-coupling has been shown to induce neural-entrainment that can synchronize walking-pace with sonic tempo. The extent to which acoustical-motor entrainment can induce longer-term changes to physical activity behaviours remains unclear.

Cardiac rehabilitation is essential and is associated with irrefutable mortality benefits for patients following an acute cardiac event. Randomized clinical trials have demonstrated a 25-50% improvement in survival as compared to controls; however, as many as 50% of patients will dropout of such programs prior to completion, which undermines these morbidity and mortality benefits (37; 54). Research exploring ways to improve compliance to such programs has suggested that the incorporation of music and other such holistic, patient-centered interventions into a rehabilitation/exercise program is associated with improved motivation, endurance and satisfaction amongst cardiac rehabilitation participants. The MAINTAIN study has been designed to conduct a feasibility evaluation on the effects of a preference-based music intervention on adherence to the cardiac rehabilitation program at Toronto Rehabilitation Institute. The primary objective of the trial is to evaluate the feasibility of the implementation of such a protocol within the context of the program.

This is a two-arm, block 2:1 randomized trial. 35 patients participating in cardiac rehabilitation at Toronto Rehabilitation: Cardiac Rehabilitation and Secondary Prevention Program will be recruited and participants will be randomized into: 1) control (standard, usual care); and, 2) music intervention. The randomization process employed will be a blocked 2:1 strategy, whereby subjects are randomized to the music treatment arms 2:1. All those patients randomized into arm 2 will be equally randomized into either (2) preference-based music intervention, (3) preference-based music enhanced with RAS. The primary outcome measure will be weekly physical activity over a 3 month duration as measured using tri-axial accelerometers. We will also analyze the impact of a preference-based music intervention based on audio playlist utilization, self-reported sitting times ,exercise-times, on-site attendance to the cardiac rehabilitation program (attendance), peak oxygen uptake (VO2) (stress-test), and self-efficacy levels (self-efficacy questionnaires). These measures will be collected and analyzed throughout the course of the intervention (3 months).

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients, who are participating in and have been declared medically stable for out-patient cardiac rehabilitation, will be recruited from the Toronto Rehabilitation Institute's Cardiac Rehabilitation and Secondary Prevention Program.

Exclusion Criteria:

* Participants who are unable to wear the MP3 device or the activity monitoring device due to medical or non-medical issues will be excluded from this study.
* Subjects that have a medical history of seizure disorders, previous neurosurgery, or known head trauma will be excluded from this study.
* Subjects that have received a bicycle-based exercise prescription.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Duration of physical activity | 3 months
  The primary outcome will be the total weekly physical activity volume as determined using triaxial accelerometers.

SECONDARY OUTCOMES:
On-site program attendance | 3 months
  Adherence will be measured quantitatively by assessing the number of missed appointments vs. amount of scheduled appointments.
Change in Cardio Pulmonary Assessment Score | Baseline, 3 months
  Fitness levels will be measured by assessing peak VO2 (ml/kg-1* min-1), an objective, clinical measure of the volume of oxygen consumed while exercising at the maximum capacity. Those with higher VO2max values are more fit and can exercise more intensely, indicating a greater functional capacity than those with lower VO2max values.
Changes in Stafford Self-Efficacy Questionnaire/Cardiac Self-Efficacy Questionnaire Scores | Baseline, 3 months
  Changes in self efficacy will be measured using the combined score of two self-efficacy questionnaires administered by Toronto Rehabilitation Institute
Audio-play list use | 3 months
  We will track the number of song plays on each patients playlist
Study recruitment and drop-out | 3 months
  We will determine the proportion of patients screened, recruited, and who completed the study protocol

OTHER OUTCOMES:
Interview and Focus Group | 3 months
  Tertiary outcomes of the study will include information gathered regarding music playlist preferences and subjective opinions about the role of music in exercise programs through post-intervention interviews (attached). Other secondary outcomes include the energy expenditure and activity time as recorded over the entire three-month period by the activity monitoring device and MP3 device (this data collected every 2 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Dr. David Alter, Principal Investigator — Toronto Rehabilitation Institute
Locations (1):
- Toronto Cardiac Rehabilitation Institute, Toronto, Ontario, Canada

REFERENCES:
- [Background] Alter DA, Iron K, Austin PC, Naylor CD; SESAMI Study Group. Socioeconomic status, service patterns, and perceptions of care among survivors of acute myocardial infarction in Canada. JAMA. 2004 Mar 3;291(9):1100-7. doi: 10.1001/jama.291.9.1100. PMID 14996779
- [Background] Chan RH, Gordon NF, Chong A, Alter DA; Socio-Economic and Acute Myocardial Infarction Investigators. Influence of socioeconomic status on lifestyle behavior modifications among survivors of acute myocardial infarction. Am J Cardiol. 2008 Dec 15;102(12):1583-8. doi: 10.1016/j.amjcard.2008.08.022. Epub 2008 Oct 9. PMID 19064009
- [Background] De Angelis C, Bunker S, Schoo A. Exploring the barriers and enablers to attendance at rural cardiac rehabilitation programs. Aust J Rural Health. 2008 Jun;16(3):137-42. doi: 10.1111/j.1440-1584.2008.00963.x. PMID 18471183
- [Background] Molloy GJ, Perkins-Porras L, Strike PC, Steptoe A. Social networks and partner stress as predictors of adherence to medication, rehabilitation attendance, and quality of life following acute coronary syndrome. Health Psychol. 2008 Jan;27(1):52-8. doi: 10.1037/0278-6133.27.1.52. PMID 18230014
- [Background] Hagan NA, Botti MA, Watts RJ. Financial, family, and social factors impacting on cardiac rehabilitation attendance. Heart Lung. 2007 Mar-Apr;36(2):105-13. doi: 10.1016/j.hrtlng.2006.05.010. PMID 17362791
- [Background] Worcester MU, Murphy BM, Mee VK, Roberts SB, Goble AJ. Cardiac rehabilitation programmes: predictors of non-attendance and drop-out. Eur J Cardiovasc Prev Rehabil. 2004 Aug;11(4):328-35. doi: 10.1097/01.hjr.0000137083.20844.54. PMID 15292767
- [Background] Glazer KM, Emery CF, Frid DJ, Banyasz RE. Psychological predictors of adherence and outcomes among patients in cardiac rehabilitation. J Cardiopulm Rehabil. 2002 Jan-Feb;22(1):40-6. doi: 10.1097/00008483-200201000-00006. PMID 11839996
- [Background] Grace SL, Gravely-Witte S, Brual J, Monette G, Suskin N, Higginson L, Alter DA, Stewart DE. Contribution of patient and physician factors to cardiac rehabilitation enrollment: a prospective multilevel study. Eur J Cardiovasc Prev Rehabil. 2008 Oct;15(5):548-56. doi: 10.1097/HJR.0b013e328305df05. PMID 18830085
- [Background] Bandura A. Health promotion by social cognitive means. Health Educ Behav. 2004 Apr;31(2):143-64. doi: 10.1177/1090198104263660. PMID 15090118
- [Background] (10) Van Noorden, L., & Moelants, D. Resonance in the perception of musical pulse. Journal of New Music Research 1999, 43-66
- [Background] van der Vlist B, Bartneck C, Maueler S. moBeat: Using interactive music to guide and motivate users during aerobic exercising. Appl Psychophysiol Biofeedback. 2011 Jun;36(2):135-45. doi: 10.1007/s10484-011-9149-y. PMID 21380562
- [Background] Konlaan BB, Bygren LO, Johansson SE. Visiting the cinema, concerts, museums or art exhibitions as determinant of survival: a Swedish fourteen-year cohort follow-up. Scand J Public Health. 2000 Sep;28(3):174-8. PMID 11045748
- [Background] Konlaan BB, Bjorby N, Bygren LO, Weissglas G, Karlsson LG, Widmark M. Attendance at cultural events and physical exercise and health: a randomized controlled study. Public Health. 2000 Sep;114(5):316-9. PMID 11035447
- [Background] Marrero DG, Fremion AS, Golden MP. Improving compliance with exercise in adolescents with insulin-dependent diabetes mellitus: results of a self-motivated home exercise program. Pediatrics. 1988 Apr;81(4):519-25. PMID 2451207
- [Background] Rhodes RE, Warburton DE, Bredin SS. Predicting the effect of interactive video bikes on exercise adherence: An efficacy trial. Psychol Health Med. 2009 Dec;14(6):631-40. doi: 10.1080/13548500903281088. PMID 20183536
- [Background] O'Konski M, Bane C, Hettinga J, Krull K. Comparative effectiveness of exercise with patterned sensory enhanced music and background music for long-term care residents. J Music Ther. 2010 Summer;47(2):120-36. doi: 10.1093/jmt/47.2.120. PMID 21141769
- [Background] Johnson G, Otto D, Clair AA. The effect of instrumental and vocal music on adherence to a physical rehabilitation exercise program with persons who are elderly. J Music Ther. 2001 Summer;38(2):82-96. doi: 10.1093/jmt/38.2.82. PMID 11469917
- [Background] Edworthy J, Waring H. The effects of music tempo and loudness level on treadmill exercise. Ergonomics. 2006 Dec 15;49(15):1597-610. doi: 10.1080/00140130600899104. PMID 17090506
- [Background] Karageorghis CI, Jones L, Priest DL, Akers RI, Clarke A, Perry JM, Reddick BT, Bishop DT, Lim HB. Revisiting the relationship between exercise heart rate and music tempo preference. Res Q Exerc Sport. 2011 Jun;82(2):274-84. doi: 10.1080/02701367.2011.10599755. PMID 21699107
- [Background] Bradt J, Dileo C. Music for stress and anxiety reduction in coronary heart disease patients. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD006577. doi: 10.1002/14651858.CD006577.pub2. PMID 19370642
- [Background] Brownley KA, McMurray RG, Hackney AC. Effects of music on physiological and affective responses to graded treadmill exercise in trained and untrained runners. Int J Psychophysiol. 1995 Apr;19(3):193-201. doi: 10.1016/0167-8760(95)00007-f. PMID 7558986
- [Background] (22) Matesic B, Cromartie F, Effects Music Has on Lap Pace, Heart Rate and Perceived Exertion Rate During a 20-Minute Self-Paced, Masters' Thesis 2011
- [Background] Everett B, Salamonson Y, Davidson PM. Bandura's exercise self-efficacy scale: validation in an Australian cardiac rehabilitation setting. Int J Nurs Stud. 2009 Jun;46(6):824-9. doi: 10.1016/j.ijnurstu.2009.01.016. Epub 2009 Mar 4. PMID 19261281
- [Background] Garatachea N, Torres Luque G, Gonzalez Gallego J. Physical activity and energy expenditure measurements using accelerometers in older adults. Nutr Hosp. 2010 Mar-Apr;25(2):224-30. PMID 20449530
- [Background] Patel SA, Benzo RP, Slivka WA, Sciurba FC. Activity monitoring and energy expenditure in COPD patients: a validation study. COPD. 2007 Jun;4(2):107-12. doi: 10.1080/15412550701246658. PMID 17530503
- [Background] Slootmaker SM, Chin A Paw MJ, Schuit AJ, van Mechelen W, Koppes LL. Concurrent validity of the PAM accelerometer relative to the MTI Actigraph using oxygen consumption as a reference. Scand J Med Sci Sports. 2009 Feb;19(1):36-43. doi: 10.1111/j.1600-0838.2007.00740.x. Epub 2008 Feb 4. PMID 18266793
- [Background] Bassett DR Jr, Ainsworth BE, Swartz AM, Strath SJ, O'Brien WL, King GA. Validity of four motion sensors in measuring moderate intensity physical activity. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S471-80. doi: 10.1097/00005768-200009001-00006. PMID 10993417
- [Background] Anshel MH, Marisi D. Effect of music and rhythm on physical performance. Res Q. 1978 May;49(2):109-13. No abstract available. PMID 725276
- [Background] Cho, Jeongmin (2009). The effect of music therapy on mood, perceived exertion, and exercise adherence of patients participating in a rehabilitative upper extremity exercise program. University of Kansas, Master's Thesis: Music Education & Music Therapy.
- [Background] Copeland BL, Franks BD. Effects of types and intensities of background music on treadmill endurance. J Sports Med Phys Fitness. 1991 Mar;31(1):100-3. PMID 1861474
- [Background] Gfeller, K. (1988). Musical components and styles preferred by young adults for aerobic fitness activities. Journal of Music Therapy, 25, 28-43.
- [Background] Hayakawa Y, Miki H, Takada K, Tanaka K. Effects of music on mood during bench stepping exercise. Percept Mot Skills. 2000 Feb;90(1):307-14. doi: 10.2466/pms.2000.90.1.307. PMID 10769915
- [Background] Karageorghis CI, Mouzourides DA, Priest DL, Sasso TA, Morrish DJ, Walley CJ. Psychophysical and ergogenic effects of synchronous music during treadmill walking. J Sport Exerc Psychol. 2009 Feb;31(1):18-36. doi: 10.1123/jsep.31.1.18. PMID 19325186
- [Background] Karageorghis, C.I., Priest, D.L., Williams, L.S., Hirani, R.M., Lannon, K.M., & Bates, B.J. (2010). Ergogenic and psychological effects of synchronous music during circuit-type exercise. Psychology of Sport and Exercise, 11, 551-559.
- [Background] Pearce, K. A. (1981). Effects of different types of music on physical strength. Perceptual and Motor Skills, 53, 351-352.
- [Background] Van Noorden, L., & Moelants, D. (1999). Resonance in the perception of musical pulse. Journal of New Music Research, 28, 43-66
- [Background] Zimmerman LM, Pierson MA, Marker J. Effects of music on patient anxiety in coronary care units. Heart Lung. 1988 Sep;17(5):560-6. PMID 3417466
- [Background] White JM. Effects of relaxing music on cardiac autonomic balance and anxiety after acute myocardial infarction. Am J Crit Care. 1999 Jul;8(4):220-30. PMID 10392221
- [Derived] Alter DA, O'Sullivan M, Oh PI, Redelmeier DA, Marzolini S, Liu R, Forhan M, Silver M, Goodman JM, Bartel LR. Synchronized personalized music audio-playlists to improve adherence to physical activity among patients participating in a structured exercise program: a proof-of-principle feasibility study. Sports Med Open. 2015;1(1):23. doi: 10.1186/s40798-015-0017-9. Epub 2015 May 8. PMID 26284164